CLINICAL TRIAL: NCT07230522
Title: Effectiveness of Hyaluronic Acid (hyaDENT BG® Gel) Compared With Enamel Matrix Proteins (Emdogain®) in the Treatment of Angular Bone Defects in Combination With a Xenograft (Bio-Oss Collagen®)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Sofia (Other)
Responsible Party: Principal Investigator, Hristina Maynalovska, Chief Assistant, Medical University of Sofia
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUS-D304-HA-EMD-001; Agreement No. D 304/18.12.2023 (Other Grant/Funding Number: Medical University of Sofia)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Periodontitis; Intrabony Periodontal Defect; Periodontal Bone Loss
Keywords: periodontal regeneration; hyaluronic acid; enamel matrix derivative; angular bone defects
MeSH Terms: conditions — Periodontitis; Alveolar Bone Loss | interventions — enamel matrix proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-Oss Collagen + HyaDent BG (Experimental): Periodontal regenerative treatment in which intrabony defects are treated with Bio-Oss® Collagen combined with HyaDent® BG (cross-linked hyaluronic acid gel). The procedure follows standard periodontal surgical protocols.
  Interventions: Biological: Bio-Oss Collagen + HyaDent BG
- Bio-Oss Collagen + Emdogain (Active Comparator): Periodontal regenerative treatment in which intrabony defects are treated with Bio-Oss® Collagen combined with Emdogain®. The procedure follows standard periodontal surgical protocols.
  Interventions: Biological: Bio-Oss Collagen + Emdogain

INTERVENTIONS:
Biological: Bio-Oss Collagen + HyaDent BG — Application of Bio-Oss® Collagen combined with HyaDent® BG (cross-linked hyaluronic acid gel) during periodontal surgery for intrabony defects. Standard regenerative protocols are followed.
  Arms: Bio-Oss Collagen + HyaDent BG
Biological: Bio-Oss Collagen + Emdogain — Application of Bio-Oss® Collagen combined with Emdogain during periodontal surgery for intrabony defects. Standard regenerative protocols are followed.
  Arms: Bio-Oss Collagen + Emdogain

SUMMARY:
The goal of this clinical trial is to learn whether hyaluronic acid (HyaDent® BG) provides similar benefits to Emdogain® when both are used with Bio-Oss® Collagen during periodontal surgery in adults with periodontal (intrabony) defects. The main questions it aims to answer are:

Does the treatment reduce probing pocket depth?

Does the treatment increase clinical attachment level?

Does the treatment increase radiographic bone fill?

Does the treatment change the gingival margin position?

Researchers will compare Bio-Oss Collagen + HyaDent BG with Bio-Oss Collagen + Emdogain to see whether HyaDent BG achieves similar improvements in clinical and radiographic outcomes as Emdogain.

Participants will:

Undergo periodontal surgery to treat the vertical bone defect(s), with either Bio-Oss Collagen + HyaDent BG or Bio-Oss Collagen + Emdogain.

Attend follow-up visits for periodontal measurements and radiographs.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 18 diagnosed with periodontal disease-Stage III or IV periodontitis;

  * Sites with bone defects and a probing pocket depth (PPD) ≥ 6 mm, accompa-nied by bleeding on probing (BoP) at re-evaluation, conducted six weeks after non-surgical periodontal therapy;
  * Full Mouth Plaque Score (FMPS) < 20% and Full Mouth Bleeding Score (FMBS) < 15% prior to surgical treatment;
  * Good general health with no systemic conditions and no known allergies to materials or medications used in the study.

Exclusion Criteria:

* Medical conditions contraindicating surgical intervention;

  * Pregnancy or lactation;
  * Heavy smokers;
  * Untreated periodontal disease;
  * Poor oral hygiene;
  * Acute infectious lesions in the area of intervention;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
periodontal pocket depth reduction | Before the surgery and 6 moths after the surgery
Clinical attachment gain | Before the surgery and 6 months after surgery
Radiographic bone fill | Before and 6 months after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Periodontology, Faculty of Dental Medicine, Medical University of Sofia, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No